Official Title of study: Assessment of Outcomes Following Bariatric Surgery for Mississippi State

Employees

NCT: 41165

Date of Document: Created April 05, 2010; uploaded May 3, 2018

Form: IRB application (study protocol and statistical analysis plan)



The University of Mississippi
Office of Research and Sponsored Programs
Division of Research Integrity and Compliance - Institutional Review Board
100 Barr Hall - University, MS 38677
irb@research.olemiss.edu

## APPLICATION TO CONDUCT RESEARCH WITH HUMAN SUBJECTS ~ Instructions ~

- Use the most recent version of this form (<a href="http://www.olemiss.edu/depts/research/compliance/compliance-forms.htm#irb">http://www.olemiss.edu/depts/research/compliance/compliance-forms.htm#irb</a>).
- Do not submit a handwritten form. Prepare as a Word document, using no less than a 10 point font. [Note that, as this is a protected form, you cannot use Spell Check. It is best to prepare text in another document first, then cut and paste.]
- Answer all of the questions on this form completely. (If you have questions about this form, please contact the DRIC office at 662-915-7482 or <a href="mailto:irb@research.olemiss.edu">irb@research.olemiss.edu</a>.)
- For examples of Abstracts, go to <a href="http://www.olemiss.edu/depts/research/compliance/human/sample\_abstracts.html">http://www.olemiss.edu/depts/research/compliance/human/sample\_abstracts.html</a>
- For examples of Procedures, go to <a href="http://www.olemiss.edu/depts/research/compliance/human/sample\_procedures.html">http://www.olemiss.edu/depts/research/compliance/human/sample\_procedures.html</a>.
- Complete and attach all supporting documentation and all appropriate appendices.
- Complete the checklist that accompanies this form to assure all requirements for submission are completed.
   Incomplete submissions will not be reviewed.
- E-mail the completed form with attachments to <u>irb@research.olemiss.edu</u>. Fax the signature page to 662-915-7577, or mail or bring it to the Office of Research and Sponsored Programs, Division of Research Integrity and Compliance, 100 Barr Hall, University, MS 38677.

CHECKLIST

| All supporting document are attached. All appropriate Approval of another community Complete copy of the graph Departmental signatures A copy of this application. List all personnel involutions. | ts (consent forms, asser<br>oriate appendices are co-<br>nmittee or another institu-<br>ant proposal, with pages<br>s (and signature of advision has been made for the<br>lived with this research | nt forms, survent forms, survent forms, survent to the control of | eys, interview q<br>attached.<br>able, is attache<br>human subject<br>research) have<br>s records.<br>ve contact wit | ts highlighted, if applicable, is attached. |
|---|---|---|---|---|
| NAME | FACULTY<br>OR STAFF | GRADUATE<br>STUDENT | UNDERGRAD<br>STUDENT | ROLE ON PROJECT |
| Katie McClendon | | | | Principal Investigator |
| Whitney Byars | | | | Oxford Surgical and Bariatric Clinic, LLC site manager |
| | | | | 04.111 |

If more space is needed to list project personnel, please submit Appendix A found on the ORSP Compliance Forms page.

OFFICE USE ONLY

## **APPLICATION TO CONDUCT RESEARCH WITH HUMAN SUBJECTS**

ABSTRACT: Briefly summarize your project using non-technical, jargon-free language that can be understood by non-scientists. Include: (1) a statement of the research question and related theory supporting the reasons for, and importance of, the research; (2) the ages and characteristics of your proposed subjects and how you will recruit them; (3) the research design; and (4) a description of the procedure(s) subjects will undergo. Limit to the space below, using no less than a 12 point font. See Instructions (page 1) for a link to examples.

- 1. Objective: to assess the health and economic outcomes (weight lost, change in control of chronic diseases such as diabetes, quality of life, work productivity, health care cost, etc) associated with bariatric (weight-loss) surgery for 200 severely obese patients who undergo bariatric surgery as part of the Mississippi State Employees' Life and Health Insurance Plan's Obesity Treatment Program (OTP).
- 2. Patient Characteristics: Inclusion criteria: Eligible bariatric surgical candidates who are enrolled in the OTP (100 patients per year for 2 years). The Plan's criteria includes, but is not limited to 1) enrollment in the plan for at least 12 consecutive months prior to September 1, 2009; 2) completion of the HealthQuotient health risk assessment through the Plan's wellness and health promotion program; 3) a Body Mass Index (BMI) of >40 kg/m2, or a BMI >35 kg/m2 with two or more co-morbidities such as diabetes, hypertension, sleep apnea or asthma; 4) two or more physician-supervised weight loss attempts within the last 24 months; 5) age 18 years or older; and 6) consent to provide personal and medical information to the Plan. Prior to surgery, each site administers a pychiatric evaluation to ensure the patient is pychologically stable for surgery. Exclusion criteria: any patient who does not meet criteria above or who declines to participate. Surgeries will take place only at Certified Bariatric Surgery Centers of Excellence (COE), of which, there are currently 3 in the state. The 3 COEs exist with 4 outpatient medical offices (1 COE is composed of 2 independent surgeon practices) Patients will be recruited at each site once they are approved by the OTP.
- 3. Design: prospective, observational, multi-center, longitudinal study of outcomes and resource utilization associated with OTP. Estimates of obesity and comorbidities' impact will be obtained from the outpatient medical office for the COEs. Medical charts, databases and medical/pharmacy claims will be the source of information. Surveys on quality of life, productivity, and patient satisfaction will be administered directly to patients. Database claim information will be obtained in future and is not a part of current IRB application.
- 4: Procedures: After obtaining informed consent, patients will be administered surveys at baseline, as well as at follow-up visits. Additional data will be obtained via patient charts, databases, and medical/pharmacy claims.

| | | Mai data min 50 optal | ned via patier | it charts, databas | res, and medicampharmacy claims. |
|---|---|---|---|---|---|
| 1. | PROJECT TITLE: Assessment of Outcomes Following Bariatric Surgery for Mississippi State Employees | | | | |
| | If student project: | dissertation | thesis 🔲 o | other: | |
| | Date dissertation or t | thesis proposal approve | ed by committe | ee: | (committee approval required) |
| 2. | PRINCIPAL INVESTIGA | ATOR: Dr. Dr. Ms. | ☐ Mr. Katie | McClendon | |
| | Department | School of Pharmacy | , Dept Pharm | acy Practice | Work Phone: 601.984.2638 |
| | Mailing Address: | 2500 North State Str | eet, Office An | nex I | Home Phone: 601.668.8811 |
| | | Jackson | MS | 39225 | 110110. 001,000,0011 |
| | E-Mail Address: | kmcclendon@sop.u | msmed.edu | | Fax Number: 601.984.2751 |
| | Co-Investigator(s) | : name | | nam | e |
| 3. | RESEARCH ADVISOR: | | - | | (required for student researchers) |
| | Department: | | | Work Phone: | |
| | E-Mail Address: | | | Fax Number: | |

| 4. | FUNDING SOURCE: | | · | | |
|---|---|---|---|---|---|
| | Is there funding for this pr | oject? X Yes | Û | External: | ding: ORSP Faculty Research Program Other: Pending/Agency: Awarded/Agency: Allergan |
| 5. | ANTICIPATED BEGINNING A<br>HUMAN SUBJECTS CONTAC | | ES OF | Beginning Date:<br>Ending Date:<br>Not Applicable: | 04/10/2010 (as soon as approved)<br>12/31/2013 |
| | 2000 Hel 1270 July 148 | RESEARC | н Метно | DOLOGY/PROC | EDURES |
| 6. | CHECK ALL PROCEDURES BE | LOW THAT APPLY | TO YOUR 5 | TUDY: | |
| - | □ Pre-existing data | <b>ਹੇ</b> ਹੈ | Ð | Source of data: | Patient medical charts, BOLD Database,<br>MS State Employee medical and<br>pharmacy claims. Claims information not<br>part of this IRB application. |
| | | | | Do data have ide | |
| | Observation Oral history Interview Focus group | | | | |
| | Questionnaire or Survey | Anonymous?<br>Distribution: | Inte | erson | Anonymous or Confidential? Anonymous means (1) the investigator cannot associate a subject with his/her data and (2) the data cannot identify a subject. Examples: Surveys with no names handed to an investigator are not anonymous; surveys placed by the subject in a group data envelope can be anonymous; surveys with no names and with demographic data that can identify a subject (e.g., the only African-American in a class) |
| | Experiment/manipulat | <b>:</b> | | | are not anonymous. |
| | ☐ Treatment study ☐ Other: | 1011 | | | |
| | ☐ Exercise ⇔ | <b>\$</b> | <b>⇔</b> | ☐ Moderate ☐ More than m | oderate |
| | ☐ Videotaping ☐ Audio recording | | | | |
| | ☐ X-rays 🗢 | <b>D D</b> | 0 | E.g. DEXA ~ conta | ct Health & Safety for training requirements. |
| | Collection/use of blood fluids, or tissues ** | <b>\$</b> | ⇔ | If Yes, has IBC a | ion been submitted? |
| | Contact Health and Safety | e <u>nttp://www.olet</u><br>for training requir | miss.edu/de<br>rements. | pis/research/comp | liance/compliance forms.html#ibc. |

| | Use of drugs, biological products, or medical devices | |
|---|---|---|
| 7. | DECEPTION OR OMISSION OF ELEMENTS OF CONSENT: Do any of the following apply to your study? The study uses surreptitious videotaping. The study gives subjects deceptive feedback, whether positive or negative. The study uses a research confederate. The study has misleading or deceptive: (1) study descriptions; (2) procedure explanations; and/or (3) survey instructions/rationales. If you checked any of the above, please complete Appendix D. | |
| | PARTICIPANT INFORMATION | |
| 8. | SUBJECT CHARACTERISTICS: Number: 200 Age Range: 18 &up | If under 18, parental consent is required. |
| 9. | BRIEFLY DESCRIBE SUBJECT POPULATION: Obese adults with state insurance | E.g. 2 <sup>nd</sup> grade students, college students, etc.<br>Justify exclusion of any racial or gender group. |
| 10. | POTENTIALLY VULNERABLE SUBJECTS INVOLVED: Children/adolescents¹ Mentally ill – outpatients Mentally ill – inpatients Cognitively impaired Elderly, if institutionalized Pregnant females Prisoners² HIV+ Other: | Check all applicable groups. <sup>1</sup> Complete Appendix B if applicable. <sup>2</sup> Complete Appendix C. |
| 11. | RECRUITMENT PROCEDURES: a. How will you recruit subjects? Check all that apply: Psych PSPM UM bulletin boards, where: Class announcements Letters to parents/guardians E-mail - specify groups: [Mass e-mails to UM groups must: 1) be in plain text; 2) state "This study has been approved by UM's Institutional Review Board (IRB); and 3) be limited to 200 words.) Radio/TV/newspaper ads Other: Patients who are approved for surgery at 4 sites as part of OTP will be enrolled. This application only pertains to Oxford Surgical & Bariatric Clinic, LLC [List all recruitment sites.] Recruitment ad/e-mail/oral announcement is attached: c. Describe incentives for subjects, if any (money, drawing, class points, etc.). | <ul> <li>b. Are subjects in a subservient power relationship to investigators or to parties with an interest in the research, such as students in an instructor/investigator's class or employees of the investigator?</li> <li>Yes No</li> <li>If Yes, how will you ensure that their participation is truly voluntary?</li> <li>Yes No</li> <li>No incentives</li> </ul> |
| | cass polits, etc.). | |

| | - | | | | |
|---|---|---|---|---|---|
| 12. | Co | NSENT PROCEDURES: Oral (attach script) Information letter – used in survey resea Informed consent form (attach) Assent form for children or subjects with (attach) | E 100 | Check all that apply. If you plan to enroll non-English participants, the consent form an document(s) must be translated appropriate language(s) and incl this submission. | d assent<br>into the<br>uded with |
| | | Not applicable Request waiver of written consent – just Request waiver of consent – justify: | ify: | For subject populations where co<br>to consent is highly questionable<br>psychiatric populations), explain<br>competency will be determined a<br>whom. | (e.g. some<br>how |
| 13. | WH | ERE WILL THE STUDY BE CONDUCTED? | | Check all that apply. | |
| | | UM campus Local community: elementary/secondar care facility <sup>1</sup> | y school(s) or child | <sup>1</sup> Complete Appendix B. | |
| | $\boxtimes$ | Local community: other - specify: 4 phy associated with 3 Certified Bariatric S Excellence in Mississippi (Jackson, O application only pertains to Oxford Su Clinic,LLC. | urgery Centers of<br>exford, Pascagoula). This | <sup>2</sup> Complete Appendix E. | |
| | | Another U.S. location – specify:<br>Another country <sup>2</sup> – specify:<br>Not applicable | | | |
| | | Approval letter from another IRB attache | ed | | |
| | | Approval letter from other organization | | | |
| 14. | DES | Physical: Patients have already | RESEARCH ASSISTANT TRA<br>emergency plan to handle | ISKS, INCLUDING EXPERIMENTER AN INING/EXPERTISE. For example, an expotential adverse events for traus schology research with children. | |
| | | chosen to receive surgery, which has risks, but this study doesn't increase risk. | | | ⊠ n/a |
| | Ъ. | Emotional: Surveys ask personal information, which may cause mild psychological stress, but no more than encountered in day-to-day life | patients could discuss v | tered at medical site, where with medical personnel. ninded that information shared | ☐ n/a |
| | c. | Social/interpersonal: Surveys ask personal information, which may cause mild psychological stress, but no more than encountered in day-to-day life | patients could discuss v | tered at medical site, where with medical personnel. ninded that information shared | n/a |
| | d. | Occupational: While subjects are employees, spouses, or retires of the State, all medical information is confidential, so there should be no occupational risk. | | | ⊠ n/a |

■ Not applicable

d. List pro-rating for incentives for study drop-outs.

| | e. | Financial: | ⊠ n/a |
|---|---|---|---|
| | f. | Legal: | ⊠ n/a |
| | g٠ | Other: | □ n/a |
| 15. | phy<br>Pati<br>wor | sical fitness, etc.) POTENTIAL BENEFITS DO NOT INCLUients who have bariatric surgery may have improve | ed health, quality of life, and improved productivity at ected to have minimal benefit to the subjects enrolled, |
| 16. | □ ⊠ □ ⊠ Wh | W WILL YOU MAINTAIN DATA CONFIDENTIALITY? All data are anonymous (go to next section). Data are confidential. Data kept in locked file cabinets. Data in locked room. en will data be de-identified? at time of lection \[ \int \n/a \] | Anonymous or Confidential? Anonymous means (1) the investigator cannot associate a subject with his/her data and (2) the data cannot identify a subject. THE IRB ENCOURAGES PERMANENT RETENTION OF DATA FOR POTENTIAL FUTURE USE BECAUSE THIS IMPROVES THE COST/BENEFIT RATIO. |

## **PROJECT DESCRIPTION**

17. DESCRIBE YOUR PROJECT IN THE SPACES BELOW.

Spaces will expand as you enter text

a. Problem statement (including specific aims of your project):

To assess the health, humanistic and economic outcomes associated with bariatric surgery for 200 severely obese patients who have State insurance and who undergo bariatric surgery as part of the Obesity Treatment Program (OTP).

b. Brief literature review that points to a need for this research:

Mississippi has the highest rate of adult obesity in the nation at 32.8% in 2008, whereas, 10 years prior, the rate was 22.8%. Obesity has far-reaching effects on the health, health care resource use, and productivity of the population. Obesity-related co-morbidities and complications include coronary artery disease (CAD), hypertension, type 2 diabetes mellitus (T2DM), cancer, non-alcoholic fatty liver disease, dyslipidemia, and sleep apnea which increase the morbidity, mortality and cost of care associated with obesity. Increases in obesity in the US population parallel a substantial share of growth in health spending and continues to impose an economic burden on both public and private payers.

Studies currently exist which evaluate the costs and benefits of bariatric surgery on an obese population, but little information is available on a population with obesity rates as high as seen in Mississippi.

Additionally, in 2009, the State of Mississippi passed legislation that authorized bariatric surgery as a covered health benefit for state employees for a select obesity program. Continued coverage past 2011 will be contingent on outcomes from the project and funding availability.

As a result of this legislation, Mississippi's State and School Employees' Life and Health Insurance Plan (SSELHI Plan) will provide a two-year Obesity Treatment Program (OTP) for the treatment and management of obesity and related conditions. Under the OTP, the Plan will provide benefits for medically necessary bariatric procedures at certified Centers of Excellence (COE) in Mississippi for qualifying participants.

c. Description of procedures:

After approval for surgery by the OTP, patients will be invited to participate in this study at the physician office associated with a COE. This application is for the Oxford Surgical & Bariatric Clinic, LLC. After completion of Consent Form, patients will be asked to fill out surveys and their providers, medical staff and/or PI will assist in filling out data collection form at initial and follow-up visits. No direct intervention to the patient will occur. Some patients have already had surgery--for these patients will have the surveys administered at next follow-up, and chart reviews will be done to fill out Initial Visit and Follow-Up Visit Data Collection Forms. Database claim information is not part of this IRB application, but will be

done in future to obtain economic outcome information.

| • | | | | | |
|----|------|-----|----|-----|----|
| d. | - N/ | 0.5 | SU | 100 | |
| • | IV. | | | | э. |

## SURVEY/TEST/QUESTIONNAIRE (e.g. WAIS)

| | CONTENT TO TO QUESTION WARE (e.g. WALD) | |
|---|---|---|
| NA | ME AND ACRONYM | IS THERE PUBLISHED PSYCHOMETRIC SUPPORT? |
| 1 | Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI: GH) | ⊠ Yes □ No |
| 2 | Impact of Weight / Quality of Life-Lite (IWQOL-Lite) | 🛛 Yes 🗌 No |
| 3 | Patient History Survey | ☐ Yes 🛛 No |
| 4 | Patient Satisfaction Survey | Yes No |
| 5 | | Yes No |
| | OTHER MEASURES (e.g. heart rate) | |
| NA | ME DEAL WAS SHEET AND SHEE | |
| 1 | Prevalence of hypertension, control of hypertension (as measured by b medication for hypertension (drug[s], dose) | elood pressure) and use of |
| 2 | Prevalence of type 2 diabetes mellitus (DM), control of DM (as measure medication for DM (drug[s], dose) | d by A1c) and use of |
| 3 | Prevalence of dyslipidemia, control of dyslipidemia (as measured by lip medication for dyslipidemia (drug[s], dose) | old levels) and use of |
| 4 | Prevalence of sleep apnea and sleep apnea score | An Jac High K I |
| 5 | Prevalence of other obesity-related complications, including but not lingastroesophageal reflux disease (GERD) and control of these diseases | nited to CAD, asthma, |
| 6. | Serum creatinine and liver function enzymes, when available in medical of | |
| 7. | Incidence of nutritional deficiencies and use of medication to treat deficie | |
| 8. | Incidence of device or surgery-related adverse events | |
| 9. | Outpatient medication costs* | |
| 10. | Hospitalization costs* | |
| 11. | Office visit costs* | |
| 12 | Emergency room costs* | |

Provide a numbered step-by-step list of all procedures, starting with recruitment. Elaborate on more complex items. Attach scripts of procedural instructions to subjects. See Instructions (page 1) for examples.

\*these items will be part of research in future and are not part of current IRB application.

- 1 Mississippi's State and School Employees' Life and Health Insurance Plan (SSELHI Plan) will determine which 200 patients will have surgery as part of the Obesity Treatment Program (OTP). 100 patients were approved in 2009, and 100 more will be approved in 2010. Patients approved for the OTP will work with the surgery team to chose the type of surgery best for the patient. Once the patient is approved for the OTP, then their participation with this study can begin.
- At the initial visit for surgery consultation, the patient will be asked if they are willing to participate in this study. If patient consents, then they will fill out the consent form with the assitance of someone at the COE (Whitney Byars). This person has been trained in admisistration of surveys by the Pl. Once the Consent Form has been signed, the patient will answer surveys (Patient History Survey, WAPI: GH, IWQOL-Lite). After this visit, medical personnel in the COE (Whitney Byars, with the assistance of the Pl when available), will fill out the Initial Visit Data Collection Form. The information for the Initial Visit Data Collection Form will come from the patient's medical record and/or the BOLD database (a database all COEs use to collect information on all surgery patients at the site).

If the patient has had surgery already, the Patient History Survey will be administered to the patient at the

next available visit.

- 3 Soon after the patient has surgery, the Peri-surgery Data Collection Form will be filled out by medical personnel at the physican's office (Whitney Byars). If needed, PI will assist in completion of this form.
- 4 At follow-up visits near 6 months, 12 months, and 24 months post-surgery at the physician office, the patient will fill out the IWQOL-lite, WPAI:GH, and Patient Satisfaction surveys. After these follow-up visits, medical personnel at the COE (with the assistance of PI when available), will fill out the Follow-up visit Data Collection Form. Information for this form will also be found in the patient chart and/or BOLD database.
- 5 If the patient has an adverse event at any time during the study, an adverse event form will be filled out by medical personnel and/or PI.
- 6. At study closure, or if patient wishes to withdraw from the study at any time, the Withdrawal/End of Study form will be filled out.
- 7. Each patient will also have a State Employee Bariatric Surgery Project Checklist, which will be filled out by Whitney Byars to ensure study methods are followed correctly.
- 8. After the patient has signed the consent form, study personnel will collaborate with CareAllies, which serves as the disease management program for the Mississippi State and School Employees' Life and Health Insurance Plan State of Mississippi. Via this collaboration, medical and pharmacy claims will be reviewed for the patient to collect information (costs) of pharmacy utilization, medical visits, emergency room visits, and hospitalizations.\* This part of the study is not a part of the current IRB application, but will be done at a later time.
- f. Data analysis methods:
  - Statistical analysis: Descriptive statistics will be reported for each measure at baseline and at the 6, 12, and 24 month followup periods. We will use a generalized linear model for repeated measurements (generalized estimating equations) to assess the effect of bariatric surgery across followup periods. This approach will also be used to assess the effect of surgery type (Roux-en-y versus banding) while controlling for the effect of other variables. An alpha of 0.05 will be used to determine statistical significance.
- g. Debriefing and/or feedback on test results (procedures, forms, scripts, and statements if applicable):

| ACCUPANCES COMMUNICATION OF LANGUAGE AND FIRST | |
|---|---|
| ASSURANCES ~ CONFLICT OF INTEREST AND FISCAL RESPONSIBIL | |
| Do you or any person responsible for the design, conduct, or reporting of this study have an e as an officer or a director of any outside entity whose financial interests may reasonably appearesearch? | conomic interest in, or act<br>ir to be affected by this |
| NO Each surgery office may have economic interest in surgery of interest in surgery o | to ensure integrity of |
| Do you or any person responsible for this study have existing financial holdings or relationshi study? | ps with the sponsor of this |
| <ul> <li>YES ⇒ ⇒ If Yes, please explain any potential conflict of interest.</li> <li>NO</li> <li>N/A</li> </ul> | |
| SIGNATURES | Talking a selection |
| PRINCIPAL INVESTIGATOR, RESEARCH ADVISOR (IF APPLICABLE) AND DEPARTMENT CHA | UR MUST SIGN BELOW |
| PRINCIPAL INVESTIGATOR'S ASSURANCE | |
| I certify that the information provided in the application is complete and correct. As Principal ultimate responsibility for the protection of the rights and welfare of the human participants, or and the ethical performance of the project. I will comply with all UM policies and procedures, applicable federal, state, and local laws regarding the protection of participants in human resellimited to the following: The research will be performed by qualified personnel according to the approved research. No changes will be made in the research protocol or informed consent document(s) until a Informed consent will be obtained from the participants, if applicable and appropriate; Adverse events and/or unanticipated problems will be reported to the IRB as required. I certify that I, and all key personnel, have completed the required initial and/or refresher CIT principles and regulatory requirements for the protection of human research participants. MCCLADIAN AMAGEMENT ASSETTION ASSETTIO | conduct of the research,<br>, as well as with all<br>arch, including, but not<br>a protocol;<br>approved by the IRB; |
| RESEARCH ADVISOR'S ASSURANCE (REQUIRED FOR STUDENT PROJECTS) As the research advisor, I certify that the student investigator is knowledgeable about the regular governing research with human participants and has sufficient training and experience to concresearch in accordance with the approved protocol. I agree to meet with the investigator on a regular basis to monitor research progress; Should problems arise during the course of the research, I agree to be available, personally investigator in solving them; I will ensure that the investigator will promptly report adverse events and/or unanticipate required; If I will be unavailable, for example, on sabbatical leave or vacation, I will arrange for an a assume responsibility during my absence and I will advise the IRB by letter or e-mail of su I have completed the required initial and/or refresher CITI courses in the ethical principle requirements for the protection of human research participants. | duct this particular t, to supervise the ed problems to the IRB as Iternate faculty member to |
| *The research advisor must be a UM faculty member. The faculty member is considered the responsit | |
| | ne party for the ethical |

| performance and regulatory compliance of the research projec | t. | |
|---|---|---|
| DEPARTMENT CHAIR'S ASSURANCE | | |
| As department chair, I acknowledge that this research is ir | keening with the standards set by | our department and I |
| certify that the Principal Investigator has met all departme | ental requirements for approval of t | his research |
| (1/10) | | - 1 1 |
| - Heide (lee 1/oss) | | 4/5/10 |
| Signature of Department Chair/Dean* | | Date |
| *If the Principal Investigator is also the department chair, this sig | nature must be that of the Dean. | |
| <u> </u> | | |
| OFFICE USE ONLY | | |
| OFFICE USE ONLY | | |
| OFFICE USE ONLY Administrative Review | | |
| Sec. | | |
| ☐ Administrative Review | | |
| ☐ Administrative Review ☐ Expedited Review: Approval expires | | |
| ☐ Administrative Review ☐ Expedited Review: Approval expires | Signature | Date |
| ☐ Administrative Review ☐ Expedited Review: Approval expires | ☐ IRB Coordinator | Date |
| ☐ Administrative Review ☐ Expedited Review: Approval expires | ☐ IRB Coordinator<br>☐ IRB Chair | Date |
| ☐ Administrative Review ☐ Expedited Review: Approval expires | ☐ IRB Coordinator | Date |

+ + + + + + ATTACH (INSERT) ADDITIONAL REQUIRED DOCUMENTS HERE + + + + + + + (all will be sent as separate documents)

| • |
|---|